CLINICAL TRIAL: NCT06182865
Title: A Prospective Study of Ga-68 Dolacga Scintigraphy to Evaluate Liver Reserve Function in Patients With Hepatocellular Carcinoma Before and After Proton Therapy
Brief Title: A Study of Ga-68 Dolacga to Evaluate Liver Reserve Function in Patients With HCC Before and After Proton Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Atomic Research Institute, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INER-V09DX-proton
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Hepatic Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ga-68 Dolacga Injection (Experimental): Ga-68 Dolacga Injection, 2.0±1.0 mCi, single dose, iv bolus
  Interventions: Drug: Ga-68 Dolacga Injection

INTERVENTIONS:
Drug: Ga-68 Dolacga Injection — Ga-68 Dolacga will be administered via iv bolus injection followed by a whole-body PET/CT scan for liver reserve evaluation.

SUMMARY:
This is a single-center, prospective, open-labeled, single-arm, interventional study to evaluate liver reserve and tumor response using Ga-68 Dolacga positron emission tomography and the safety of the investigational product in patients with hepatocellular carcinoma before and after proton therapy.

DETAILED DESCRIPTION:
This is a single-center, prospective, open-labeled, single-arm, interventional study to evaluate liver reserve and tumor response using Ga-68 Dolacga positron emission tomography and the safety of the investigational product in patients with hepatocellular carcinoma before and after proton therapy.

This trial will enroll 10 eligible subjects. All subjects will provide informed consent before any study procedures are performed. Screening procedures (visit 1) will occur within 21 days prior to imaging visit (visit 2) and will include: inclusion/exclusion criteria check, pregnancy test (if applicable), vital signs, laboratory tests, electrocardiogram (ECG) and establishment of baseline characteristics. Primovist MRI will occur within 14 days prior to imaging visit (visit 2) and 1 week after imaging visit (visit 4), and will be performed according to standard procedure of study site.

The baseline characteristics include medical/medication history, fibrosis index, Child-Pugh score and classification, MELD score, liver oncology diagnosis, tumor size, preoperative treatments (portal vein embolization, transarterial chemoembolization, transarterial embolization or biliary drainage), existence of thrombosis (portal vein thrombosis or hepatic vein thrombosis). The liver tissue fibrosis index FIB-4 will be measured to assess the morphological changes.

During the imaging session (visit 2, Day 1; visit 4, Day 84±3), a catheter will be placed for intravenous (IV) administration of Ga-68 Dolacga. Subjects will receive an iv bolus injection of 2.0±1.0 mCi Ga-68 Dolacga. A PET/CT scan will be kinetically performed for 60 minutes immediately after IV injection.

The measurement of liver reserve is the primary endpoints of this study and measurement will be evaluated by Ga-68 Dolacga PET. The measurement of liver reserve will be performed at visit 2 and visit 4 of this study for all subjects. Adverse events will be continuously monitored during the imaging session.

Two follow-up visits (visit 3 at Day 7±2 and visit 5 at Day 91±2) will be conducted to confirm subject well-being and to collect information about any new adverse events (if any).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hepatocellular carcinoma and scheduled to have the PBT.
* 20~80 years old
* Performance status: ECOG 0-1
* Child-Pugh class A

Exclusion Criteria:

* Massive or uncontrolled ascites
* Concurrent with other malignancy
* Under pregnancy or breastfeeding
* With distant metastasis
* Allergic to investigational drug(s) or similar drug(s)/ formulation(s);
* Known hypersensitivity to PRIMOVIST
* Acute or chronic severe renal insufficiency (glomerular filtration rate <30 mL/min/1.73m^2)
* General PET and MRI exclusion criteria
* Can't follow our follow-up schedule because of any reason

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of liver reserve obtained from the Ga-68 Dolacga PET performed in HCC patients before proton therapy. | Visit 2 (Day 1)
  The liver reserve parameters obtained from Ga-68 Dolacga PET is expressed in "percentage of injection dose (%ID) and standard uptake value, (SUV)."
Measurement of liver reserve obtained from the Ga-68 Dolacga PET performed in HCC patients after proton therapy. | Visit 4 (Day 84±3)
  The liver reserve parameters obtained from Ga-68 Dolacga PET is expressed in "percentage of injection dose (%ID) and standard uptake value, (SUV)."

SECONDARY OUTCOMES:
Number of subjects with clinically significant changes in systolic blood pressure and diastolic blood pressure | from pre-dose to visit 2 (Day 1), visit 3 (Day 7±2), visit 4 (84±3), and visit 5 (Day 91±2)
Number of subjects with body temperature abnormalities | from pre-dose to visit 2 (Day 1), visit 3 (Day 7±2), visit 4 (84±3), and visit 5 (Day 91±2)
Number of subjects with clinically significant changes in Heart Rate | from pre-dose to visit 2 (Day 1), visit 3 (Day 7±2), visit 4 (84±3), and visit 5 (Day 91±2)
Number of subjects reporting clinically significant changes in serum biochemical tests | from pre-dose to visit 2 (Day 1), visit 3 (Day 7±2), visit 4 (84±3), and visit 5 (Day 91±2)
Number of subjects reporting clinically significant changes in hematological tests | from pre-dose to visit 2 (Day 1), visit 3 (Day 7±2), visit 4 (84±3), and visit 5 (Day 91±2)
Number of subjects reporting clinically significant changes in urinalysis | from pre-dose to visit 2 (Day 1), visit 3 (Day 7±2), visit 4 (84±3), and visit 5 (Day 91±2)
Number of subjects with clinically significant changes in electrocardiogram(ECG) | from pre-dose to visit 2 (Day 1), visit 3 (Day 7±2), visit 4 (84±3), and visit 5 (Day 91±2)
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 91 days
  All laboratory abnormalities which are compared with screening values and out of the reference range will be considered as AE and will be assessed its relationship to the study drug. Any ECG changes including ECG waveform will be assessed as AE(s) and will be followed to assess whether they resolved and when they resolved.

CONTACTS AND LOCATIONS:
Overall Officials: Bing-Shen Huang, MD, Principal Investigator — Linkon Chang Gung Memorial Hospital
Locations (1):
- Linkon Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No